CLINICAL TRIAL: NCT01159093
Title: Using Health Information Technology to Improve Healthcare Quality in Primary Care Practices and in Transitions Between Care Settings
Brief Title: Giving Immunizations Through Vaccine Education
Acronym: GIVE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 09-00-7352; AHRQ (Other Grant/Funding Number: HHSA29032001T)
Record Dates: First submitted 2010-07-07; First posted 2010-07-09 (Estimated); Last update posted 2015-03-12 (Estimated); Status verified 2011-08

CONDITIONS: HPV Vaccines
Keywords: Clinical Decision Support Systems

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Family Decision Support (Experimental): Families will receive informational vaccine reminder telephone calls.
  Interventions: Behavioral: Family Decision Support
- Clinical Decision Support (Experimental): In this treatment arm, clinicians receive the decision support at the point of care within an electronic health record.
  Interventions: Behavioral: Clinician Decision Support
- Family DS+ Clinician DS (Experimental): Families will receive informational vaccine reminder calls and their clinicians will receive electronic health record-based decision support for immunizations.
  Interventions: Behavioral: Family Decision Support; Behavioral: Clinician Decision Support; Other: Family Decision Support and Clinician Decision Support
- Control (Other): This group will receive regular primary care with no decision support.
  Interventions: Other: Control

INTERVENTIONS:
Behavioral: Family Decision Support — Family-focused intervention includes informational vaccine reminder telephone calls prompted by an electronic health record.
  Other Names: Clinical Decision Support; Family Focused Intervention
  Arms: Family DS+ Clinician DS; Family Decision Support
Behavioral: Clinician Decision Support — Clinician-focused intervention includes an electronic health record-based decision support mechanism including reminders, education, audit and feedback on vaccination success.
  Other Names: Clinical Decision Support; Clinician Focused Intervention
  Arms: Clinical Decision Support; Family DS+ Clinician DS
Other: Family Decision Support and Clinician Decision Support — This will be a combination of the family-focused decision support (telephone reminder calls) and clinician-focused decision support (clinical alerts).
  Other Names: Family Decision Support; Clinician Decision Support
  Arms: Family DS+ Clinician DS
Other: Control — Usual care
  Arms: Control

SUMMARY:
This study will test the effectiveness of clinician-focused health IT-based decision support, family-focused health IT-based decision support, and a combination of both efforts, in increasing HPV and other adolescent vaccine rates among adolescent girls. We hypothesize that a combination of clinician-focused clinical decision support and family-focused decision support will be most effective.

DETAILED DESCRIPTION:
* Clinician-focused intervention includes an electronic health record-based decision support mechanism including reminders, education, audit and feedback on vaccination success.
* Family-focused intervention includes vaccine reminders and informational telephone calls prompted by the electronic health record.

ELIGIBILITY:
Inclusion Criteria:

* All clinicians practicing at participating sites
* Parents with an eligible adolescent girl
* Adolescent girls
* Ages 11-17
* Has a visit at one of the primary care centers within the last 15 months.
* Has not completed the teen vaccine series

Exclusion Criteria:

* None

Ages: 11 Years to 17 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child
Enrollment: 23675 (Actual)
Dates: Start 2010-05; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Rate of HPV vaccination among girls actively cared for at participating sites | Monthly, up to 1 year
  The outcome will be assessed monthly, until study completion (1 year).

SECONDARY OUTCOMES:
Rates of meningococcal and tetanus, diphtheria, and pertussis vaccines among girls in the study | Monthly, up to 1 year
  The outcome will be assessed monthly, until study completion (1 year).

CONTACTS AND LOCATIONS:
Overall Officials: Alexander G Fiks, MD, MSCE, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Mayne SL, duRivage NE, Feemster KA, Localio AR, Grundmeier RW, Fiks AG. Effect of decision support on missed opportunities for human papillomavirus vaccination. Am J Prev Med. 2014 Dec;47(6):734-44. doi: 10.1016/j.amepre.2014.08.010. Epub 2014 Nov 18. PMID 25455116